CLINICAL TRIAL: NCT06021678
Title: A Phase I/II Study Evaluating the Safety, Efficacy, and Pharmacokinetics of EX103 in Subjects with Relapsed/Refractory CD20-Positive Non-Hodgkin Lymphoma
Brief Title: Safety and Efficacy of EX103 in Subjects with Relapsed/Refractory CD20-Positive Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Excelmab Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EX103-001
Record Dates: First submitted 2023-08-22; First posted 2023-09-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: CD20-positive Non-Hodgkin Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EX103 injection (Experimental): From Cycle 0 to Cycle 2, the subject will receive the preset dose of EX103 once a week (QW), and from Cycle 3, the subject will receive the preset dose of EX103 once every two weeks (Q2W). The recommended dose is MTD or OBD, and a cycle of treatment is 28 days.
  Interventions: Drug: EX103 injection

INTERVENTIONS:
Drug: EX103 injection — Administered as specified in the treatment arm.
  Other Names: EX103; bispecific monoclonal antibody that recognizes both CD3 and CD20

SUMMARY:
This is a multicenter, single-arm, open, dose-escalation Phase I/II clinical trial, consisting of a dose-escalation phase (accelerated titration phase, 3+3 design) and a dose expansion phase.

DETAILED DESCRIPTION:
Based on the safety, tolerability, PK results, and antitumor activity of EX103 in patients with relapsed or refractory CD20-positive non-Hodgkin lymphoma, this study will determine dose-limiting toxicity (DLT) and determine the maximum tolerated dose (MTD) or optimal biological dose (OBD) to provide a basis for the recommended Phase 2 dose (RP2D). The dose expansion phase will further evaluate the safety, tolerability, PK, PD profile, initial antitumor effect, and immunogenicity of several extended cohorts.

ELIGIBILITY:
Inclusion Criteria:

-

1. Provision of signed and dated informed consent form; stated willingness to comply with all study procedures and availability for the duration of the study; 2. Aged ≥ 18 years old, male or female; 3. Meeting the following criteria:

1. Dose-escalation phase: (1) with CD20-positive non-Hodgkin lymphoma confirmed at the first diagnosis (excluding patients whose CD20 turned negative after rituximab treatment); (2) with relapsed or refractory disease after least 2 prior lines of systemic therapy; (3) currently with no suitable therapy available for prolonging survival;
2. Dose-expansion phase:

(i) Cohort 1:

1. Histopathologically and immunohistochemically confirmed CD20-positive diffuse large B-cell lymphoma (DLBCL) (excluding patients whose CD20 turned negative after rituximab treatment) : including non-specific (NOS) DLBCL, high-grade B-cell lymphoma (HGBCL), primary mediastinal (thymus) large B-cell lymphoma (PMBCL), and translational follicular lymphoma (trFL) (patients who have converted from follicular lymphoma to DLBCL can be enrolled, and pathology reports should be provided at the same time if there is a disease transformation), or follicular lymphoma (FL) with histological grade 3b; the sponsor may limit the number of patients with PMBCL and trFL enrolled;
2. Previous failure or relapse after second-line or higher systemic treatment regimens (at least one of which included anti-CD20 targeted therapy and at least one of which included anthracyclines);

(ii) Cohort 2:

1. Histopathologically and immunohistochemically confirmed CD20-positive follicular lymphoma (FL) (excluding patients whose CD20 turned negative after rituximab treatment);
2. The histological grade ranged from 1 to 3a;
3. Previous failure or recurrence of second-line or higher systemic regimens (at least one of which included anti-CD20 targeted therapies and alkylating agents; The sponsor may limit the minimum number of patients who are refractory to both anti-CD20-targeted therapies and alkylating agents);
4. Must be indicative of treatment due to symptoms and/or tumor burden;

(iii) Cohort 3:

1. Histopathologically and immunohistochemically confirmed CD20-positive non-Hodgkin lymphoma (excluding patients with CD20 turning negative after rituximab treatment), other than the types included in cohort 1 and cohort 2; the sponsor may limit the number of patients with certain or several specific tumor species to be enrolled;
2. Previous failure or relapse after second-line or higher standard treatment, at least one of which included a combination of anti-CD20 monoclonal antibodies and chemotherapy agents;
3. In cases of indolent lymphoma, indications for treatment must be present due to symptoms and/or tumor burden;

4. At the dose escalation and expansion stages, the subjects must have at least one two- dimensionally measurable lesion as the basis for evaluation by CT, or MRI, if CT is not applicable: for intranodal lesions, the long diameter is ≥ 1.5 cm; for extranodal lesions, the long diameter is ≥ 1.0 cm;

5. ECOG performance status score: 0-2;

6. Life expectancy ≥ 12 weeks;

7. The laboratory test results should be met before each cycle beyond cycle 1 (blood components, short-acting cell growth factors, albumin, and other drugs are not allowed to be given within the first 7 days of laboratory tests; long-acting cell growth factors are not allowed to be given within the first 14 days):

1. Absolute neutrophil count ≥ 1.0×109/L;
2. Platelet count ≥ 50×109/L;
3. Hemoglobin ≥ 80 g/L;
4. Serum total bilirubin ≤ 1.5×ULN; if there is liver invasion, serum total bilirubin ≤ 3×ULN;
5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; if there is liver invasion, ALT and AST ≤ 5×ULN;
6. Serum creatinine ≤1.5×ULN or creatinine clearance estimated by Cockcroft-Gault formula ≥ 30 mL/min;
7. International normalized ratio (INR) or plasma prothrombin time (PT) ≤ 1.5×ULN;

   8. Women of childbearing potential and men with a partner of childbearing potential who consent to use highly effective methods of birth control during treatment and for an additional 90 days after the last administration of the protocol specified treatment; women of childbearing age without surgical sterilization must have a negative result in serum HCG test within 7 days before enrollment in the study and isn't breastfeeding.

   Exclusion Criteria:
   1. Clear history of drug allergy, foreign protein, biologics or ingredients of investigational drugs;
   2. Uncontrolled active infection during the screening period;
   3. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplant; or received autologous hematopoietic stem cell transplantation (HSCT) or CAR-T cell therapy within 3 months;
   4. CNS metastases, or other serious central nervous system diseases (such as epilepsy, cerebral infarction, and cerebral hemorrhage) within 6 months, History of neurodegenerative condition or CNS movement disorder. Subjects with a history seizure within 12 months prior to study enrollment are excluded;
   5. At least one active person is known to have human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Subjects with evidence below are eligible for study entry:

      1. Human immunodeficiency virus antibody (HIV-Ab) is negative;
      2. Hepatitis B surface antigen (HBsAg) is negative; when HbsAg or HbcAb is positive, HBV-DNA (HBV deoxyribonucleic acid) is < lower limit of detection;
      3. Hepatitis C virus antibody is positive, and HCV RNA is negative.
   6. Toxicities caused by previous anti-tumor therapy has not recovered to grade ≤ 1 (CTCAE v5.0), except alopecia and other tolerable events as determined by the investigator;
   7. Develop any other malignancy within 5 years (except for completely treated cervical carcinoma in situ or basal cell or squamous cell skin cancer);
   8. Use of any vaccine within 4 weeks prior to initial pretreatment with dexamethasone or methylprednisolone or during the intended study period;
   9. Systemic immunosuppressive drugs, including but not limited to radiotherapy immune conjugate, antibody drug conjugations, immune/cytokines, monoclonal antibodies, etc., have been used within 4 weeks prior to initial pretreatment with dexamethasone or methylprednisolone.
   10. With a history of active autoimmune diseases, including but not limited to myocarditis, pneumonia, myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, multiple sclerosis, vasculitis, or glomerulonephritis;
   11. Any condition that the investigator believes may not be appropriate for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) [dose escalation (Cycle 0 and Cycle 1)] | During the DLT evaluation period (28 days from Cycle1 Day1 at the dose escalation stage).
  To determine the RP2D and the MTD, if reached.
Safety endpoints：incidence and severity of adverse events (AE), laboratory tests, etc. | From first dose until the end of the safety follow-up period [within 28 ± 7 days after the last study treatment or before the start of other anti-tumor treatments (whichever occurs earlier)].
  Treatment-emergent AEs (TEAEs) as assessed by CTCAE v5.0. Abnormal laboratory values are reported as AEs per protocol.

SECONDARY OUTCOMES:
All parts: Time to reach Cmax (Tmax) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Tmax is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Maximum (peak) plasma concentration (Cmax) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Cmax is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Area under the concentration-time curve from time 0 to the last measurable concentration using linear-log trapezoidal rule (AUC0-t) | From first dose until treatment discontinuation, expected average of 3.5 years.
  AUC0-t is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Elimination half-life (t 1/2) | From first dose until treatment discontinuation, expected average of 3.5 years.
  t 1/2 is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Total body clearance of drug from the plasma (CL) | From first dose until treatment discontinuation, expected average of 3.5 years.
  CL is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Steady-state maximum plasma concentration(Css,max) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Css,max is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Steady-state minimum plasma concentration(Css,min) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Css,min is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Steady-state time to maximum concentration(Tss,max) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Tss,max is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Area under the plasma concentration versus time curve at Steady-State(AUCss) | From first dose until treatment discontinuation, expected average of 3.5 years.
  AUCss is one of the characteristics of Pharmacokinetic (PK) endpoint.
All parts: Pharmacodynamic (PD) endpoint | From first dose until treatment discontinuation, expected average of 3.5 years.
  Before and after administration of EX103, changes in lymphocyte subsets and peripheral blood cytokine levels.
All parts: Objective response rate (ORR) | From first dose until treatment discontinuation, expected average of 3.5 years.
  ORR is defined as the proportion of subjects whose optimal response is CR or CRi or PR. Subjects who did not undergo tumor evaluation after baseline were considered to have no objective, as determined by the investigator using Lugano 2014 criteria.
All parts: Disease control rate (DCR) | From first dose until treatment discontinuation, expected average of 3.5 years.
  DCR is defined as the proportion of subjects whose best response is CR or CRi or PR or SD.
All parts: Duration of response (DoR) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Duration of response (DoR) is defined as the time between the first onset of CR or CRi or PR and the onset of PD or death from any cause, whichever occurs first, in subjects with objective response.
All parts: Incidence of anti-drug antibodies (ADA) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Percentage of positive patients of anti-drug antibody.
All parts: Incidence of neutralizing antibody (NAb) | From first dose until treatment discontinuation, expected average of 3.5 years.
  Percentage of positive patients of neutralizing antibody.
All parts: Confirmation of anti-drug antibody and neutralizing antibodies. | From first dose until treatment discontinuation, expected average of 3.5 years.
  Screening of antibodies against corresponding antigens and confirmation of positive antibodies, and determination of the titers of related antibodies (IgG, etc.) produced in the humoral and cellular immunity.

CONTACTS AND LOCATIONS:
Overall Officials: Junyuan Qi, MD, PHD, Principal Investigator — Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - Cancer Hospital Affiliated to Zhengzhou University, Henan Cancer Hospital, Zhengzhou, Henan
  - Qilu Hospital, Cheeloo College of Medicine, Shandong University, Jinan, Shandong
  - Shanghai Sixth People's Hospital, Shanghai Jiaotong University school of Medicine, Shanghai, Shanghai Municipality
  - Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality